CLINICAL TRIAL: NCT06531278
Title: Adebelimab Combined With Irinotecan Liposomal Injection, Oxaliplatin, Fluorouracil and Calcium Folinate Are Used in the First-line Treatment of Pancreatic Cancer Liver Metastasis Efficacy and Safety
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiang Long (Other)
Responsible Party: Sponsor-Investigator, Jiang Long, Chief physician of hepatobiliary and pancreatic surgery, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MR-31-24-025345
Record Dates: First submitted 2024-07-18; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Pancreatic Cancer Metastatic to Liver
MeSH Terms: interventions — irinotecan sucrosofate; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- first-line treatment of pancreatic cancer liver metastasis efficacy and safety (Experimental): Adebelimab combined with irinotecan liposomal injection, oxaliplatin, Fluorouracil and calcium folinate
  Interventions: Drug: Irinotecan liposome; Drug: Adebrelimab; Drug: Oxaliplatin; Drug: Fluorouracil; Drug: Calcium folinate

INTERVENTIONS:
Drug: Irinotecan liposome — * Patients are planned to receive irinotecan liposomal (60 mg/m2; d1) of every cycle.
  * 27 days a cycle
Drug: Adebrelimab — * Patients are planned to receive Adebrelimab (20 mg/kg; d1) of every cycle.
  * 27 days a cycle
Drug: Oxaliplatin — * Patients are planned to receive Oxaliplatin (85 mg/m2; d1) of every cycle.
  * 27 days a cycle
Drug: Fluorouracil — * Patients are planned to receive fluorouracil (2400mg/m2; d1) of every cycle.
  * 27 days a cycle
Drug: Calcium folinate — * Patients are planned to receive Calcium folinate (400mg/m2; d1) of every cycle.
  * 27 days a cycle

SUMMARY:
1. Evaluation of adebelimab in combination with irinotecan liposomes, oxaliplatin, fluorouracil, efficacy and safety of leucovorin in the first-line treatment of advanced metastatic pancreatic cancer
2. Construct the model of immunotherapy combined with chemotherapy for the treatment of pancreatic cancer liver metastasis

DETAILED DESCRIPTION:
Pancreatic cancer is a cancer of the digestive system with a very high degree of malignancy and a very poor prognosis. In recent years, morbidity and death. The rate shows a clear upward trend at home and abroad. Global cancer statistics in 2020 show that there are new pancreas cases worldwide each year. There are about 495,000 cases of adenocarcinoma and about 466,000 deaths from pancreatic cancer each year. Statistical tables for 2020. In the United States, there are about 57,600 new cases of pancreatic cancer every year, and about 47,050 deaths due to pancreatic cancer each year. Data from pancreatic cancer collected by the National Cancer Center of China in 2019. show that the incidence of pancreatic cancer in Chinese is:6.92 per 100,000, with new cases accounting for about 4.31% of all malignant tumors; The case fatality rate is 6.16 per 100,000 and deaths per year Cases account for about 3.78% of all malignancies. The specific etiology and pathogenesis of pancreatic cancer are unclear, and most (85%). It is an adenocarcinoma originating from the ductal epithelium. Early symptoms are atypical, and most patients are diagnosed locally advanced or out. Now distant metastasis. In the past decade, the first-line treatment regimen for pancreatic cancer has been AG, FOLFIRINOX, GS as the commonly used chemotherapy regimens, and the median OS was 8.5 months, 11.1 months, and 10.1 months, respectively. First-line treatment for pancreatic cancer still needs to be explored. The advent of plastid Iriconia has changed the landscape of first-line treatments, and the NAPOLI-3 study compared NALIRINOX (liposome irinotecan, oxaliplatin, fluorouracil, leucovorin) and AG regimens in the first-line treatment of metastatic pancreatic cancer and safety, with a median follow-up of 16.1 months, showed that the median OS of NALIRINOX versus AG was respectively 11.1 versus 9.2 months (HR 0.83 [95% CI 0.70-0.99]; p=0.036), and the median PFS was 7.4 vs. 5.6, respectively months (HR 0.69 [0.58-0.83]; p<0.0001), the ORR was 42% and 36%, respectively. Based on this research The FDA approved liposomal irinotecan in combination with oxaliplatin, fluorouracil, and leucovorin for the first-line treatment of metastatic pancreas Indications for adenocarcinoma.

Jiangsu Hengrui Pharmaceutical Co., Ltd. developed irinotecan hydrochloride liposome injection (HR070803) has both protection Protective, long-term cyclic and passively targeted. HR070803 combination with 5-FU/LV for second-line treatment of locally advanced or metastatic pancreas after failure of gemcitabine therapy Adenocarcinoma. Significantly prolonged the subject's OS compared to placebo in combination with 5-FU/LV, with a clinically meaningful difference, Significantly lower risk of death. In addition, HR070803 in combination with 5-FU/LV may also prolong the subject's PFS and TTF, and improve ORR and CA19-9 response rates. At the same time, HR070803 combined with 5-FU/LV in advanced pancreas. The type of AE observed in the treatment of adenocarcinoma is consistent with that of regular irinotecan, and there are gastrointestinal reactions, hematotoxic. It is less sexual, well tolerated, and safe and controllable.

Based on the above evidence, this study explored the efficacy and safety of adebelimab, irinotecan liposome, oxaliplatin, fluorouracil, and leucovorin in the first-line treatment of advanced metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily join this study and sign the informed consent form
2. Age: 18-75 years old (inclusive), male or female
3. Histologically confirmed pancreatic cancer liver metastases and no previous treatment of any systemic anti-swelling tumor treatment
4. No central nervous system metastases
5. No adjuvant therapy within 6 months prior to enrollment
6. ECOG PS: 0~1 points
7. Estimated survival ≥ 12 weeks
8. Normal function of major organs, meeting the following requirements (7 prior to initiation of study treatment days): (1) Routine blood examination: (No blood transfusion and no use of granules within 14 days before screening.) Cell colony-stimulating factor [G-CSF], not corrected with medication):1) Hemoglobin [HB]≥90g/L; 2) Absolute neutrophil count [ANC] ≥1.5×10 9 /L； 3) Platelets [PLT] ≥80×10 9 /L； (2) Blood biochemistry tests must meet the following criteria (no transfusion in the 14 days before screening Protein): 1) Serum total bilirubin [TBIL] ≤ 1.5 times the upper limit of normal (ULN); 2) Alanine aminotransferase [ALT], aspartate aminotransferase [AST]<2.5×ULN ； If there is liver metastasis, ALT and AST≤5×ULN； 3) Blood creatinine [Cr]≤1×ULN or endogenous creatinine clearance rate > 50ml/min (Cockcroft-Gault formula); (3) International normalized ratio [INR] ≤ 2.3 or prothrombin time [PT] exceeding Over the range of normal controls≤6 seconds: (4) Urine protein < 2+ (if urine protein ≥ 2+, you can urinate eggs for 24 hours White quantitative, 24-hour urine protein quantification <1.0g can be enrolled);
9. Women of childbearing potential must have a pregnancy test (serum or urine) within 7 days prior to enrollment The result is negative and voluntarily during the observation period and after the last dose of study drug8 Use of appropriate methods of contraception within a week; For males, it should be surgically sterile, or Agrees to adopt appropriate during the observation period and for 8 weeks after the last dose of study drug method contraception
10. Those who are expected to have good compliance can follow up the efficacy and adverse reactions according to the requirements of the protocol.

Exclusion Criteria:

1. Other active malignancies within 5 years or concomitantly
2. Have uncontrolled cardiac clinical symptoms or diseases, such as: (1) in accordance with: New York Heart Association (NYHA) criteria grade II or greater cardiac insufficiency or Cardiac ultrasonography: LVEF (left ventricular ejection fraction) <50%; (2) Instability Stereotyped angina; (3) Myocardial infarction within 1 year prior to the start of study treatment Die; (4) Clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention: (5) QTc>450ms (male); QTc>470ms (Women) (The QTc interval is calculated by Fridericia's formula; If the QTc is abnormal, interval can be used Approximately 2 minutes for three consecutive tests, taking the average);
3. Those who have high blood pressure and cannot be reduced to the normal range by antihypertensive drug treatment (admitted Systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg) (based on 2 measurements of ≥ The mean of the BP readings obtained), which is allowed to be achieved through the use of antihypertensive therapy above parameters
4. Coagulation abnormalities (INR>1.5×ULN, APTT>1.5×ULN), with: Bleeding tendency
5. Active bleeding
6. Uncontrolled active infection, chronic infectious disease, immunodeficiency syndrome
7. Subjects with known active hepatitis B (HBsAg positive and HBV DNA ≥10 3 copy number or ≥1000 U/ml)
8. Presence of active autoimmune disease or history of autoimmune disease with possible recurrence 9. Known history of severe allergy to the study drug
9. Uncontrolled infection at screening
10. Other patients who are considered by the treating physician to be unsuitable for inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | Up to 1 year after the treatment
  The proportion of patients whose tumors shrink to a certain amount for a certain period of time and include cases of complete response (CR) and partial response (PR). Calculated as: (CR cases + PR cases) / FAS × 100 (%); FAS (full analysis set) refers to the case of qualified patients, administered more than one case.
  Tumor remission rates are calculated according to the RECIST guidelines (version 1.1)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China